CLINICAL TRIAL: NCT05996029
Title: A Joint Real-World Study of Digital Smoking Cessation Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Hangzhou Medisol Technology Co. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: K4011
Record Dates: First submitted 2023-07-31; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-05

CONDITIONS: Tobacco Smoke Pollution; Passive Smoking; Secondhand Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intensive intervention package "Quit with Love" (1 month)
  1. Cognitive-behavioral (CBT) smoking cessation intervention
  2. ACT cessation intervention with positive thinking
  3. Online group smoking cessation intervention through live streaming
  "Quit Assistant" intelligent support platform (3 months)
  1. Quit smoking punch card toolkit
  2. Machine learning algorithm-driven cessation assistance practice service
  Interventions: Combination Product: Digital Smoking Cessation
- control group (No Intervention): Reduced functionality of the Love Quit applet Only a simple smoking punch card support function, mainly used to assist subjects to quit smoking on their own and collect follow-up information

INTERVENTIONS:
Combination Product: Digital Smoking Cessation — The core technology of the study is a smoking cessation assistance practice service driven by a machine learning algorithm. The small programs used by the intervention group in this study included smoking cessation service packages based on cognitive behavioral therapy and online guidance from medical staff on staff, and more digital smoking cessation tools.
  Arms: Intervention group

SUMMARY:
According to the "China Smoking Health Hazard Report 2020", the total number of smokers in China is estimated to be 350 million, of which 180 million are already addicted. In addition, more than 700 million nonsmokers are exposed to secondhand smoke and become passive smoking victims, among which the family is one of the main places of secondhand smoke exposure, and mothers and children are the most affected group.

Passive smoking is a risk factor for spontaneous abortion in pregnant women and an important risk factor for the occurrence of gestational hypertension syndrome and pregnancy complications, and it also affects embryonic development with adverse pregnancy outcomes such as miscarriage, stillbirth, intrauterine growth retardation, preterm birth, immune deficiency, birth defects, and mental retardation.

Helping smokers quit is the fundamental solution to reducing secondhand smoke exposure. The accessibility and effectiveness of traditional offline smoking cessation intervention services do not meet the needs of society. With the development of mobile communication technology, digital cessation such as SMS cessation, WeChat cessation, and APP cessation have emerged, which combine clinical cessation guidelines with software technology and present rich product features and interactive design, providing a new solution to expand the accessibility of clinical cessation interventions and address the problem of secondhand smoke exposure.We hope to explore the impact of different digital cessation tools and their combinations on reducing smoking prevalence and maternal tobacco exposure.

DETAILED DESCRIPTION:
This project is a two-arm, practical-utility randomized controlled trial.The study was designed to enroll 2214 quitters, and maternal cessation of enrollment after completion of the quitter enrollment.After self-reported exposure to secondhand smoke has been tested with a free cotinine urine test and the pregnant woman has signed an informed consent, she invites the smoker who is causing her secondhand smoke to quit, which may include her husband, family, friends, colleagues, neighbors, etc., or the pregnant woman herself.

Invited smokers will choose a quit day within two weeks of enrollment, use a cognitive behavioral therapy-based cessation package and online coaching from medical staff, as well as additional digital cessation tools, and receive a 12-week follow-up (smoking/quit status). Enrolled pregnant women will receive general education on maternal and child health management and the dangers of tobacco, and will be encouraged to provide psychological support and encouragement to invited quitters in the mini-program (provided both parties volunteer). The pregnant women will receive a 16-week follow-up (secondhand smoke exposure).

At the end of the study, all pregnant women and those who self-report successful cessation will receive a free cotinine test as an objective test of cessation effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women's inclusion criteria A. Adult females during gestation and within 42 days after delivery B. I do not smoke, but I self-reported secondhand smoke exposure problems
2. Inclusion criteria for smoking quitters A. Adults over the age of 18 who smoke every day; B. I have a clear intention to quit smoking;

Exclusion Criteria:

1. Maternal maternal exclusion criteria A. I am a smoker (pregnant women who are willing to quit smoking can join the smoking cessation group) B. Self-report had no risk of secondhand smoke exposure
2. Exclusion criteria for smoking quitters A. Receiving other smoking cessation interventions; B. having a severe mental illness or psychological disorder C. No smart phone or not skilled to use WeChat mini program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2214 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Biologically validated subject withdrawal rate | through study completion, an average of 4 months
  Urine cotinine concentrations was determined using a cotinine test kit (colloidal gold) at the end of follow-up.
Biologically validated maternal environmental tobacco exposure rate | through study completion, an average of 4 months
  Urine cotinine concentration was determined using a cotinine test kit (colloidal gold method) at the end of enrollment and follow-up to determine the exposure of second-hand smoke.

SECONDARY OUTCOMES:
Engagement and adherence to digital smoking cessation interventions | through study completion, an average of 4 months
  Actual enrollment and enrollment of invited participants in the digital cessation population.
  Proportion of subjects in the intervention group who completed a digital cessation intervention session.
Self-reported abstinence rates for subjects at weeks 1, 2, 3, 4, 8, and 12 after quitting date | through study completion, an average of 4 months
Changes in maternal and smoking cessation subjects' respective psychological scale assessments at baseline and at the end of follow-up | through study completion, an average of 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of ob gyn, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No